CLINICAL TRIAL: NCT00793832
Title: The Effect of Supervised Cardiorespiratory Endurance Exercise Training on Physical Fitness and Energy Expenditure in Roun-en-Y Gastric Bypass and Gastric Banding Surgery Patients.
Brief Title: The Effect of Supervised Exercise on Physical Fitness and Energy Expenditure in Post Bariatric Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Abhimanyu Garg, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCRC 837
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2010-01

CONDITIONS: Post-bariatric Surgery
Keywords: weight loss
MeSH Terms: conditions — Weight Loss | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Supervised exercise.
  Interventions: Behavioral: supervised exercise
- 2 (Active Comparator): Diet Advice
  Interventions: Behavioral: Diet advice

INTERVENTIONS:
Behavioral: supervised exercise — supervised exercise
  Arms: 1
Behavioral: Diet advice — Diet Advice
  Arms: 2

SUMMARY:
It is hypothesized that the patients in the EXDA group will be able to complete a structured exercise program at a level sufficient to accumulate at least 2000 kcal per week, and that the structured endurance activity will increase their physical fitness and total daily energy expenditure compared to the DA group.

ELIGIBILITY:
Inclusion Criteria:

1. RYGB or GB surgery patients who are at least 12 weeks post surgery
2. BMI of 40 or more
3. age 18-70years
4. sedentary lifestyle (energy expenditure of <35 kcal/kg/day measured by 7-day physical activity recall and no regular moderate physical activity exceeding 20 min/day within the previous 3 months)
5. willingness to alter physical activity in accordance with the intervention programs
6. English or Spanish speaking.

Exclusion Criteria:

1. body weight > 180 kg
2. cardiovascular disease
3. pulmonary disease
4. uncontrolled hypertension (resting DBP >100 or SBP >180 mm of Hg)
5. visual or hearing impairment
6. functional limitations (difficulty walking one-quarter mile or climbing 10 stairs)
7. abnormal ECG on VO2max test ( >1 mm ST segment depression at < 5 METS or with symptoms such as atrial fibrillation, complex ventricular arrhythmias and 3rd degree atrioventricular block)
8. known liver disease due to causes other than nonalcoholic steatohepatitis (liver transaminases > 2.5 times the upper limits of normal [SGPT>105 U/L, SGPT>120 U/L] or total bilirubin >1.5 mg/dL)
9. hematocrit of less than 30%
10. current alcohol abuse (>7 drinks or 210 g/wk for women and >14 drinks or 420 g/wk for men)
11. recreational drug abuse
12. current use of any drugs capable of inducing weight loss (e.g., orlistat, sibutramine, topiramate, etc.)
13. major neuro-psychiatric illnesses impeding competence or compliance
14. pregnancy and lactation
15. chronic renal insufficiency (serum creatinine > 2 mg/dL)
16. untreated thyroid disorders such as hypothyroidism and hyperthyroidism; and 17) bariatric surgical complications including anastomotic leak, wound complications, thrombotic disorders, intestinal obstruction, stomal complications, GI bleeding, recurrent severe abdominal pain, bilious vomiting.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Exercise at a level sufficient to accumulate at least 2000kcal per week | 12 weeks

SECONDARY OUTCOMES:
To compare body weight and composition, quality of life, fasting lipids and lipoproteins, and glycemic control between the two groups. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Meena Shah, Ph.D, Principal Investigator — University of Texas Southwestern Medical Center